CLINICAL TRIAL: NCT05665270
Title: A Randomized, Controlled Study to Evaluate the Safety and Effectiveness of Treatment
Brief Title: A Study for Post op Inflammation After Cataract Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Wyse Eyecare (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WCG IRB Protocol #20225859
Record Dates: First submitted 2022-11-10; First posted 2022-12-27 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract | interventions — Calcium Dobesilate

STUDY DESIGN:
Intervention Model Description: This is a randomized, controlled study to assess the safety and effectiveness of treatment with an intracanalicular dexamethasone (0.4mg) insert when utilized in conjunction with topical steroids as part of an extended taper steroid regimen following cataract surgery in patients with a history of epiretinal membrane, diabetic retinopathy, or non-exudative macular degeneration Group 1 (20 eyes) will receive treatment with topical 1% Prednisolone Acetate drops QID x 1 week, then Dextenza will be inserted at the one-week postoperative evaluation (Day 8).
  Group 2 (20 eyes) will receive treatment with topical 1% Prednisolone Acetate for five weeks with dosing schedule: QID x 2 weeks, TID x 1 week, BID x 1 week, QD x 1 week.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dextenza (Experimental): Group 1 (20 eyes) will receive treatment with topical 1% Prednisolone Acetate drops QID x 1 week, then Dextenza will be inserted at the one-week postoperative evaluation (Day 8).
  Interventions: Drug: Dextenza 0.4Mg Ophthalmic Insert
- Prednisolone Acetate (Active Comparator): Group 2 (20 eyes) will receive treatment with topical 1% Prednisolone Acetate for five weeks with dosing schedule: QID x 2 weeks, TID x 1 week, BID x 1 week, QD x 1 week.
  Interventions: Drug: Prednisolone Acetate 1%

INTERVENTIONS:
Drug: Dextenza 0.4Mg Ophthalmic Insert — Group 1 (20 eyes) will receive treatment with topical 1% Prednisolone Acetate drops QID x 1 week, then Dextenza will be inserted at the one-week postoperative evaluation (Day 8). Both groups will receive topical Prolensa Qa.m. x 5 weeks and Moxifloxacin TID x 1 week, per investigators preferential treatment regimen.
  Arms: Dextenza
Drug: Prednisolone Acetate 1% — Group 2 (20 eyes) will receive treatment with topical 1% Prednisolone Acetate for five weeks with dosing schedule: QID x 2 weeks, TID x 1 week, BID x 1 week, QD x 1 week.
  Both groups will receive topical Prolensa Qa.m. x 5 weeks and Moxifloxacin TID x 1 week, per investigators preferential treatment regimen.
  Arms: Prednisolone Acetate

SUMMARY:
This is a randomized, controlled study to assess the safety and effectiveness of treatment with an intracanalicular dexamethasone (0.4mg) insert when utilized in conjunction with topical steroids as part of an extended taper steroid regimen following cataract surgery in patients with a history of epiretinal membrane, diabetic retinopathy, or non-exudative macular degeneration.

DETAILED DESCRIPTION:
There will be approximately 40 eyes with two groups:

Group 1 (20 eyes) will receive treatment with topical 1% Prednisolone Acetate drops QID x 1 week, then Dextenza will be inserted at the one-week postoperative evaluation (Day 8).

Group 2 (20 eyes) will receive treatment with topical 1% Prednisolone Acetate for five weeks with dosing schedule: QID x 2 weeks, TID x 1 week, BID x 1 week, QD x 1 week.

Both groups will receive topical Prolensa Qa.m. x 5 weeks and Moxifloxacin TID x 1 week, per investigators preferential treatment regimen.

Each subject's participation is expected to last for approximately 5 weeks and subjects will be required to complete six scheduled visits over the course of the study period: Baseline (Screening Visit Day -1), Operative Visit (Day 0), Day 1, Day 8 (insertion day), Day 14, and Day 37.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be eligible for study participation if they:

1. Are planning to undergo non-complicated CCI CE/PCIOL in one or both eyes and have a history of epiretinal membrane, diabetic retinopathy, or non-exudative macular degeneration.
2. Are willing and able to comply with clinic visits and study related procedures
3. Are willing and able to sign the informed consent form
4. Patients age 18yo+

Exclusion Criteria:

Subjects are not eligible for study participation if they:

1. Have active infectious systemic disease
2. Have active infectious ocular or extraocular disease
3. Have an obstructed nasolacrimal duct in the study eye(s) (dacryocystitis)
4. Have known hypersensitivity to dexamethasone or are a known steroid responder
5. Have a history of ocular inflammation or macular edema
6. Are currently being treated with immunomodulating agents in the study eye(s)
7. Are currently being treated with immunosuppressants and/or oral steroids
8. Are currently being treated with corticosteroid implant (i.e. Ozurdex)
9. Have a history of herpes simplex virus keratitis or present active bacterial, viral, or fungal keratitis in either eye
10. Have a history of complete punctal occlusion in one or both punctum
11. Currently use topical ophthalmic steroid medications
12. Are currently pregnant or nursing.
13. Are unwilling or unable to comply with the study protocol
14. Are determined by the Investigator to not be included for reasons not already specified (e.g., systemic, behavioral, or other ocular disease/abnormality) or if the health of the subject or the validity of the study outcomes may be compromised by the subject's enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-01-30 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
Absence of anterior chamber cells | at Day 14
  SUN Scale (0 minimum/better to 4 maximum/ worse)

SECONDARY OUTCOMES:
BCVA | Baseline (day 8) to day 37
  Snellen Chart
Number of subjects requiring rescue steroid | Day 8 to Day 37
  Addition of steroid treatment
Number and Percentage of subjects with complete absence of cell | Day 8 to 37
  SUN Scale
Measuring Cell | Day 8, 14, 37
  Sun Scale (0 minimum/better to 4 maximum/ worse)
Measuring Flare | Day 8, 14, 37
  Sun Scale (0 minimum/better to 4 maximum/ worse)
Eye Pain | Day 8, 14, 37
  VAS Questionnaire 0 no pain to 10 worst possible pain
Ease of insertion | Day 8
  Noted as Easy, Moderate, or Difficult
Ease of Visualization | Day 8, 14, 37
  Noted as Easy, Moderate, or Difficult
Number of attempts to successfully insertion | Day 8
  Note Number of attempts to successfully insert as 1,2,3 attempts
Dry Eye | Day 8, Day 14, and Day 37.
  SPEED Survey Lower score indicates less dryness which is better than a higher score
Central Macular Thickness | Baseline to Day 37
  Mean change of Central Macular Thickness by Optical coherence tomography
Insert Retention | Day 8 to 37 days
  By slit lamp exam if insert is visualized or not

CONTACTS AND LOCATIONS:
Locations (1):
- Wyse Eyecare, Northbrook, Illinois, United States

IPD SHARING:
Plan to Share IPD: No